CLINICAL TRIAL: NCT06634264
Title: Comparison of Two Reeducation Methods in Children With Persistent Sleep Apnea, a Randomized Controlled Trial
Acronym: PERSIST-B-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nelly Huynh, Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A00-M09-24B (23-12-087)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea of Child; Sleep-Disordered Breathing; Adenotonsillar Hypertrophy
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Children with a sleep study positive for Obstructive Sleep Apnea would be randomized in the intervention arm (flexible oral appliance) or control group (nasal hygiene). They will be followed in parallel groups for 3 months before another sleep study/clinical examination (pre surgical) and once again after surgery ( post surgical sleep study/clinical examination).
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The sleep technician grading the sleep studies would be blind from the group, The ENT surgeons/treating physicians would be blinded from the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Soft Oral Appliance) (Experimental): Parents and participants will be instructed in wearing the soft/flexible oral appliance and how to perform nasal hygiene in order to better tolerate the device. The oral appliance comes in several sizes, adapted to the age of the child; it is constructed in a soft elastomer material, in a position of slight propulsion and opening of the mandible to help clear the pharynx. It has a ramp to guide the tongue in a good position, a labial screen to stretch the labial strap and prevent the tongue from protruding between front teeth.
  Interventions: Device: Soft Oral Appliance
- Control Arm (Nasal Hygiene) (No Intervention): Parents and Participants of this group will be reminded the nasal hygiene procedures (depending on the site; for example application of saline in each nostril three times a day,few simple breathing exercises), and given a diary to report daily use.

INTERVENTIONS:
Device: Soft Oral Appliance — Ora-Motor training of oral muscles (tongue, lips) associated with nasal hygiene, with reduced parental support.
  Other Names: Passive Oral Myofunctional Therapy with soft oral appliance; Oral Trainer
  Arms: Intervention Arm (Soft Oral Appliance)

SUMMARY:
Myofunctional therapy has been shown to be effectively reduce symptoms of paediatric obstructive sleep apnea, usually performed after adenotonsillectomy.

This study aims to evaluate the effectiveness of Passive Oral Myofunctional Reeducation (using a flexible oral appliance) compared to nasal hygiene alone (control group), in a population of children scheduled for adenotonsillectomy.

DETAILED DESCRIPTION:
Paediatric Obstructive Sleep Apnea (PedOSA) is a multifactorial condition, associated with significant comorbidities, affecting cardiovascular health, cognitive development and quality of life. Its main cause is adenotonsillar hypertrophy, but some co-factors such as obesity, orofacial dysfunctions and craniofacial abnormalities contribute to the severity of symptoms or their persistance after adeno-tonsillectomy.

Aim : Myofunctional therapy has been shown to reduce Apnea-Hyponea indexes (AHI) of children, and can serve as an adjunct to other therapies, but the level of compliance is a limiting factor. The investigator's aim is to evaluate the effectiveness of Passive Oral Myofunctional Reeducation (a flexible oral appliance) in a group a children scheduled for adeno-tonsillectomy (in association with nasal hygiene) and to compare them with nasal hygiene alone (control group).

Methods : The design of the study is a randomized Controlled Trial, enrolling 60 children with significant obstructive sleep apnea and divided into 2 groups : Group 1 using of a flexible oral appliance during quiet activities and sleep (+nasal hygiene), and Group 2 using nasal hygiene alone (control group). The objective assessment of sleep parameters is performed at home using an ambulatory device (AHI, desaturation index, minimal oxygen saturation, flow limitation, snoring), before and after therapy, in a 3-month interval. An orthodontic and craniofacial assessment, the examination of orofacial functions and tongue/lip strength measurements (IOPI system), as well as quality of life questionnaires (OSA-18) are also performed on participants, before and after therapy.

ELIGIBILITY:
Inclusion Criteria:

participants must:

* present signs of obstructive sleep apnea: snoring, apnea / respiratory pauses audible by the entourage (objectivized by a score, to the Pediatric Sleep Questionnaire (PSQ) , greater than or equal to 0.33- This questionnaire comprises twenty-two Questions and has a good sensitivity (83%) and specificity (87%) in screening for pediatric sleep apnea.
* be programmed for adenoidectomy, tonsillectomy or adeno-tonsillectomy within 3 months (or more).

Exclusion Criteria:

participants should not:

* present with a craniofacial syndrome nor a severe medical condition with complex medical management,
* present with an abnormality of the neuromuscular tone (such as Duchenne myopathy or cerebral palsy)
* receive orthodontic therapy during the study
* have a class III malocclusion (mandibular prognathy type), for which a propulsion oral appliance is contraindicated because it may aggravate mandibular prominence. Maxillary deficiency is not a exclusion criterion.
* A non-nutritive oral habit such as digital sucking (or pacifier) that persists because it interferes with oral reeducation and is a contraindication to orthodontic treatments. Children who have recently stopped such a habit may be included in the study.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Parameters Changes : Respiratory Events Index per hour (REI) and Obstructive REI | Baseline, after 3 months of intervention, then 3 months after surgery
  Full Night Polygraph using an ambulatory device Type III (cardio-respiratory); measurement of the index of apnea and hypopnea/ in relation to total sleep time, according the American Association of Sleep Medicine (AASM) recommandations for children.
Sleep Parameters Changes : Oxygen desaturation index (ODI) | Baseline, after 3 months of intervention, then 3 months after surgery
  Full Night Polygraph using an ambulatory device Type III (cardio-respiratory); measurement of the index of oxygen desaturation per hour/ in relation to total sleep time, according the American Association of Sleep Medicine (AASM) recommandations for children (oximetry).
Sleep Parameters Changes : Flow Limitation index | Baseline, after 3 months of intervention, then 3 months after surgery
  Full Night Polygraph using an ambulatory device Type III (cardio-respiratory); measurement of flow limitations per hour , in relation to total sleep time, according the American Association of Sleep Medicine (AASM) recommandations for children (nasal canula or thermistance).

SECONDARY OUTCOMES:
Oral muscles strength | Baseline, after 3 months of intervention, then 3 months after surgery
  Lip and Tongue strength and endurance measurement with the IOPI measurement system: Measurement of Anterior and Posterior tongue elevation strength (kPa), Lip Seal strength (kPa)
Reported quality of life | Baseline, after 3 months of intervention, then 3 months after surgery
  OSA 18 Questionnaire, consisting of a 18-items score and Visual Analog scale (from 0 to 10), filled by parents.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Huynh, PhD, Principal Investigator — St. Justine's Hospital; Julia Cohen-Levy, DDSMscPhD, Principal Investigator — McGill University
Locations (1):
- CHU Sainte Justine, Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided